CLINICAL TRIAL: NCT04164966
Title: Development of Novel Biomarkers for the Early Diagnosis of Type 1 Diabetes
Acronym: HONEY
Status: Active, not recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1459977
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New onset Type 1 Diabetes
- Healthy Normal Volunteers (HNV)

SUMMARY:
The purpose of this study is to measure the levels of certain substances (biomarkers) in the body that may indicate the triggers of Type 1 Diabetes, to find a better way to diagnose the disease, as well as to follow its progression.

ELIGIBILITY:
Inclusion Criteria:

Type 1 Diabetes (T1D)

1. Age 12-18 years inclusive
2. Diagnosis of T1D according to American Diabetes Association (ADA) criteria with an acute onset and presence of islet associated autoantibody by history.
3. T1D duration of ≤ 3 months from the diagnosis

Healthy Normal Volunteers (HNV)

1. Age 12-18 years inclusive
2. No personal history of diabetes according to ADA criteria
3. No history of T1D or insulin treated diabetes in first degree relatives (FDR)

Exclusion Criteria:

Acute or chronic medical conditions or medication that would contraindicate the participation in the research testing or could potentially affect metabolic and immune function including, but not limited to:

1. History of type 2 diabetes
2. Suspicion of non-type 1 diabetes (e.g. maturity onset diabetes of the young or secondary diabetes)
3. History of thyroid dysfunction in which the participant has not been on a stable dose (at least 6 weeks prior to enrollment) of thyroid replacement medication or antithyroid drugs.
4. History of cancer within the last 5 years (skin cancers, with the exception of melanoma, may be acceptable).
5. History of organ transplant
6. History of HIV, active Hepatitis B or C, or Tuberculosis
7. Pregnancy, lactation or 6 months postpartum from the scheduled date of collection
8. Psychiatric disease prohibiting adherence to study protocol
9. Use of oral or injectable anti-hyperglycemic agents: metformin, sulfonylureas, DPP-4 inhibitors, SGLT2 inhibitors, thiazolidinediones, acarbose, GLP-1 analogs.
10. Use of any other medications known to influence glucose, fat and/or energy metabolism within the last 3 months (e.g., growth hormone therapy, glucocorticoids [steroids], prescribed medications for weight loss, etc.)
11. Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete study visits

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Males and females 12-18 years of age with a diagnosis of type 1 diabetes within the past 3 months or those who do not have diabetes.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Characterization of circulating β cell-specific exosomes in children with T1D and healthy normal controls using baseline samples | 2-3 hours
  Measure will be the number (concentration) of circulating beta-cell specific exosomes. If the characterization of circulating beta-cell specific exosomes is not feasible in children with T1D due to the potentially limited low input amount of this type of exosomes in the circulation of these participants, an alternative analysis will be implemented.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pratley, MD, Principal Investigator — Study principal investigator
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Imperatore G, Boyle JP, Thompson TJ, Case D, Dabelea D, Hamman RF, Lawrence JM, Liese AD, Liu LL, Mayer-Davis EJ, Rodriguez BL, Standiford D; SEARCH for Diabetes in Youth Study Group. Projections of type 1 and type 2 diabetes burden in the U.S. population aged <20 years through 2050: dynamic modeling of incidence, mortality, and population growth. Diabetes Care. 2012 Dec;35(12):2515-20. doi: 10.2337/dc12-0669. PMID 23173134
- [Background] Dabelea D, Mayer-Davis EJ, Saydah S, Imperatore G, Linder B, Divers J, Bell R, Badaru A, Talton JW, Crume T, Liese AD, Merchant AT, Lawrence JM, Reynolds K, Dolan L, Liu LL, Hamman RF; SEARCH for Diabetes in Youth Study. Prevalence of type 1 and type 2 diabetes among children and adolescents from 2001 to 2009. JAMA. 2014 May 7;311(17):1778-86. doi: 10.1001/jama.2014.3201. PMID 24794371
- [Background] Nathan DM; DCCT/EDIC Research Group. The diabetes control and complications trial/epidemiology of diabetes interventions and complications study at 30 years: overview. Diabetes Care. 2014;37(1):9-16. doi: 10.2337/dc13-2112. PMID 24356592
- [Background] Deshpande AD, Harris-Hayes M, Schootman M. Epidemiology of diabetes and diabetes-related complications. Phys Ther. 2008 Nov;88(11):1254-64. doi: 10.2522/ptj.20080020. Epub 2008 Sep 18. PMID 18801858
- [Background] Skyler JS, Greenbaum CJ, Lachin JM, Leschek E, Rafkin-Mervis L, Savage P, Spain L; Type 1 Diabetes TrialNet Study Group. Type 1 Diabetes TrialNet--an international collaborative clinical trials network. Ann N Y Acad Sci. 2008 Dec;1150:14-24. doi: 10.1196/annals.1447.054. PMID 19120262
- [Background] Jacobsen LM, Haller MJ, Schatz DA. Understanding Pre-Type 1 Diabetes: The Key to Prevention. Front Endocrinol (Lausanne). 2018 Mar 6;9:70. doi: 10.3389/fendo.2018.00070. eCollection 2018. PMID 29559955
- [Background] Freeman DW, Noren Hooten N, Eitan E, Green J, Mode NA, Bodogai M, Zhang Y, Lehrmann E, Zonderman AB, Biragyn A, Egan J, Becker KG, Mattson MP, Ejiogu N, Evans MK. Altered Extracellular Vesicle Concentration, Cargo, and Function in Diabetes. Diabetes. 2018 Nov;67(11):2377-2388. doi: 10.2337/db17-1308. Epub 2018 May 2. PMID 29720498
- [Background] Sims EK, Evans-Molina C, Tersey SA, Eizirik DL, Mirmira RG. Biomarkers of islet beta cell stress and death in type 1 diabetes. Diabetologia. 2018 Nov;61(11):2259-2265. doi: 10.1007/s00125-018-4712-1. Epub 2018 Aug 15. PMID 30112687
- [Background] Garcia-Contreras M, Shah SH, Tamayo A, Robbins PD, Golberg RB, Mendez AJ, Ricordi C. Plasma-derived exosome characterization reveals a distinct microRNA signature in long duration Type 1 diabetes. Sci Rep. 2017 Jul 20;7(1):5998. doi: 10.1038/s41598-017-05787-y. PMID 28729721
- [Background] Robbins PD, Dorronsoro A, Booker CN. Regulation of chronic inflammatory and immune processes by extracellular vesicles. J Clin Invest. 2016 Apr 1;126(4):1173-80. doi: 10.1172/JCI81131. Epub 2016 Apr 1. PMID 27035808
- [Background] Ying W, Riopel M, Bandyopadhyay G, Dong Y, Birmingham A, Seo JB, Ofrecio JM, Wollam J, Hernandez-Carretero A, Fu W, Li P, Olefsky JM. Adipose Tissue Macrophage-Derived Exosomal miRNAs Can Modulate In Vivo and In Vitro Insulin Sensitivity. Cell. 2017 Oct 5;171(2):372-384.e12. doi: 10.1016/j.cell.2017.08.035. Epub 2017 Sep 21. PMID 28942920
- [Background] Thery C, Zitvogel L, Amigorena S. Exosomes: composition, biogenesis and function. Nat Rev Immunol. 2002 Aug;2(8):569-79. doi: 10.1038/nri855. No abstract available. PMID 12154376
- [Background] Cianciaruso C, Phelps EA, Pasquier M, Hamelin R, Demurtas D, Alibashe Ahmed M, Piemonti L, Hirosue S, Swartz MA, De Palma M, Hubbell JA, Baekkeskov S. Primary Human and Rat beta-Cells Release the Intracellular Autoantigens GAD65, IA-2, and Proinsulin in Exosomes Together With Cytokine-Induced Enhancers of Immunity. Diabetes. 2017 Feb;66(2):460-473. doi: 10.2337/db16-0671. Epub 2016 Nov 21. PMID 27872147
- [Background] Koliha N, Wiencek Y, Heider U, Jungst C, Kladt N, Krauthauser S, Johnston IC, Bosio A, Schauss A, Wild S. A novel multiplex bead-based platform highlights the diversity of extracellular vesicles. J Extracell Vesicles. 2016 Feb 19;5:29975. doi: 10.3402/jev.v5.29975. eCollection 2016. PMID 26901056
- [Background] Seyhan AA, Nunez Lopez YO, Xie H, Yi F, Mathews C, Pasarica M, Pratley RE. Pancreas-enriched miRNAs are altered in the circulation of subjects with diabetes: a pilot cross-sectional study. Sci Rep. 2016 Aug 25;6:31479. doi: 10.1038/srep31479. PMID 27558530
- [Background] Nunez Lopez YO, Retnakaran R, Zinman B, Pratley RE, Seyhan AA. Predicting and understanding the response to short-term intensive insulin therapy in people with early type 2 diabetes. Mol Metab. 2019 Feb;20:63-78. doi: 10.1016/j.molmet.2018.11.003. Epub 2018 Nov 16. PMID 30503831
- [Background] Nunez Lopez YO, Pittas AG, Pratley RE, Seyhan AA. Circulating levels of miR-7, miR-152 and miR-192 respond to vitamin D supplementation in adults with prediabetes and correlate with improvements in glycemic control. J Nutr Biochem. 2017 Nov;49:117-122. doi: 10.1016/j.jnutbio.2017.08.007. Epub 2017 Aug 26. PMID 28945992
- [Background] Korutla L, Rickels MR, Hu RW, Freas A, Reddy S, Habertheuer A, Harmon J, Korutla V, Ram C, Naji A, Vallabhajosyula P. Noninvasive diagnosis of recurrent autoimmune type 1 diabetes after islet cell transplantation. Am J Transplant. 2019 Jun;19(6):1852-1858. doi: 10.1111/ajt.15322. Epub 2019 Mar 18. PMID 30801971
- [Background] Lundberg RL, Marino KR, Jasrotia A, Maranda LS, Barton BA, Alonso LC, Nwosu BU. Partial clinical remission in type 1 diabetes: a comparison of the accuracy of total daily dose of insulin of <0.3 units/kg/day to the gold standard insulin-dose adjusted hemoglobin A1c of </=9 for the detection of partial clinical remission. J Pediatr Endocrinol Metab. 2017 Aug 28;30(8):823-830. doi: 10.1515/jpem-2017-0019. PMID 28753540
- See also: Website for AdventHealth Translational Research Institute — https://www.adventhealthresearchinstitute.com/research/translational-research-metabolism-diabetes